CLINICAL TRIAL: NCT00284791
Title: Lamotrigine Use in Treatment Refractory Depression in Adolescents
Brief Title: Lamotrigine in Treatment Resistant Depression in Adolescents
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: MaineHealth (Other)
Collaborators: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MMC-2571
Record Dates: First submitted 2006-01-30; First posted 2006-02-01 (Estimated); Last update posted 2017-05-17 (Actual); Status verified 2017-05

CONDITIONS: Adolescent Depression
MeSH Terms: interventions — Lamotrigine; Pharmaceutical Preparations; Fluoxetine; Sertraline

INTERVENTIONS:
Drug: Lamotrigine (drug)
Drug: Fluoxetine (drug)
Drug: sertraline (drug)

SUMMARY:
The primary hypothesis of this study is that in fluoxetine (Prozac)-resistant adolescents with Major Depressive Disorder (MDD), Lamotrigine plus fluoxetine will be safe and as effective as sertraline (Zoloft).

Our Primary Aim is to determine the efficacy and safety of Lamotrigine-augmentation of fluoxetine for treatment-resistant depression in adolescents.

Our Secondary Aims are to characterize the factors associated with treatment-resistance for adolescents with major depression. Also to assess the relationships in the families of adolescents with major depression as they enter treatment, and to track the differences in family relationships for adolescents who respond or do not respond. We postulate that tense, frustrated, irritable, and over-involved relationships constitute a risk factor for attenuated improvement or relapse.

DETAILED DESCRIPTION:
Mood disorders in youth, which include Major Depressive Disorder (MDD) and Bipolar Disorder (BPD), are highly prevalent, and are associated with significant mortality and morbidity. Many youths with major depression fail first-line treatments with psychotherapy and psychotropic medications. Lamotrigine (Lamictal®) recently gained approval by the FDA for maintenance treatment of bipolar disorder in adults. A few pilot studies have also shown promising results for lamotrigine (LTG) in treatment refractory mood disorders in both youth and adults, especially for depressive symptoms (Carandang et al., 2003; Frye et al., 2000).

For this proposed study, the modified design begins with adolescents with major depressive disorder who have not responded to a trial of a selective serotonin reuptake inhibitor antidepressant (SSRI), fluoxetine, of adequate dose and duration, and randomizes them either to a second SSRI or to fluoxetine augmented by lamotrigine. Non-responders to 8 weeks of fluoxetine, on at least 40 mg/day, who have not had to discontinue fluoxetine because of adverse effects, would be randomized to: (A) continue fluoxetine with lamotrigine augmentation, for 8 weeks, as in the active arm of the original Stage 2, or (B) discontinue fluoxetine and begin a second SSRI, for 8 weeks. We will use sertraline as the second SSRI, because of the data supporting efficacy from the randomized placebo-controlled trial by Wagner, et.al. (JAMA, '03). Citalopram is also a possibility (Wagner et.al, Am J. Psychiatry '04), but it has been in use for a shorter period of time than sertraline.

To maintain the blind, the B group will receive placebo augmentation.

The assessments and outcome measures would be the same as in the original study. We will consult with primary care offices to coach them through doing the initial, Stage 1, fluoxetine trial in their offices, and we will monitor the progress of adolescents started on fluoxetine in our clinic. Consent will be discussed only with those who are not responding, and treatment in the study will involve only the post-randomization treatment.

Background

Mood disorders in youth are common and debilitating. Early-onset of mood disorders often indicates a severe illness, with high likelihood of recurrence into adulthood. For prepubertal children, point prevalence of MDD is 2%, and 6% in adolescents, while the lifetime prevalence for MDD in adolescents is 20% (Birmaher et al., 2002). The duration of a Major Depressive Episode in youth ranges from 3 to 9 months, with 10% lasting more than 2 years, 60-70% recurring in adulthood, and 20-40% developing Bipolar Disorder within 5 years (Weller and Weller, 2000). The prevalence of prepubertal bipolar disorder is estimated at 0.5%. Prevalence of bipolar disorder in adolescents is 1% (Lewinshon et al., 1995). Suicide is the third leading cause of death in the 15 - 24 year old age group (10.1 per 100,000) and the fifth leading cause in the 5 - 14 year old group (0.7 per 100,00), and is highly correlated with MDD and BPD (Pfeffer, 2002). In addition, mood disorders in youth can impair functioning, often characterized by poor school performance, impaired relationships, delinquent behavior, and substance abuse.

ELIGIBILITY:
Inclusion Criteria:

1. Adolescents (13-17) diagnosed with a major depressive episode (MDE) (DSM-IV criteria) from either major depressive disorder (MDD) or bipolar disorder (BPD). BPD can present as a major depressive episode, with previous or subsequent cycling into a hypomanic, manic, or mixed episode. By definition, major depressive disorder MDD requires the presence of a major depressive episode, without cycling into a hypomanic, manic, or mixed episode.
2. CDRS (Children's Depression Rating Scale) > 40.
3. CGAS (Children's Global Assessment Scale) < 60.

   * Exclusion Criteria:

Adolescents who meet the following criteria will be excluded from the study:

1. Prior medically serious suicide attempt, within 3 months of enrollment into study or a score of 3 on suicide questions within KSADS at initial visit or the side effect checklist on follow up visits regarding current state.
2. Known or suspected mental retardation. For patients with known mental retardation, full scale IQ below 70 should be documented.
3. Current significant physical illnesses (e.g. diabetes mellitus, asthma, cystic fibrosis, congenital heart defects, genetic disorders). Patients with seizure disorders taking anticonvulsants will be excluded (no concomitant anticonvulsants).
4. Current drug or alcohol abuse. No active abuse will be permitted within two weeks of beginning the study trial (confirmed by urine testing in all cases of suspected abuse).
5. Females who are sexually active and are unwilling or considered unable to use appropriate contraception.
6. Use of benzodiazepines and other anxiolytics, antipsychotic medications, other antidepressants, stimulant medication, other mood stabilizers (e.g., lithium, valproate), and other sedative-hypnotics will not be permitted

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50
Dates: Start 2006-01 (Actual); Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas R Robbins, MD, Principal Investigator — Maine Medical Center Psychiatry Department; William McFarlane, MD, Study Director — Maine Medical Center, Center for Psychiatric Research
Locations (1):
- Maine Medical Center Outpatient Psychiatry, Portland, Maine, United States